CLINICAL TRIAL: NCT04542460
Title: Chronic Total Coronary Occlusion; Arrhythmia in Patients With Adjunction of PCI to Optimal Medical Treatment Versus Optimal Medical Treatment and in Patients With Failed PCI.
Brief Title: The Nordic Baltic Chronic Total Occlusion (CTO) Arrhythmia Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Leif Thuesen (Other)
Responsible Party: Sponsor-Investigator, Leif Thuesen, Head of PCI Research, Aalborg University Hospital
Organization: Aalborg University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CTO-ARRHYTHMIA
Record Dates: First submitted 2020-09-03; First posted 2020-09-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Chronic Total Coronary Occlusion

STUDY DESIGN:
Intervention Model Description: Investigator conceived, initiated and driven 1:1 randomized open label clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Optimal Medical Treatment (No Intervention): CTO patients receiving optimal medical treatment
- Optimal Medical Treatment and PCI (Active Comparator): CTO patients receiving PCI in ajunction to optimal medical treatment
  Interventions: Procedure: PCI

INTERVENTIONS:
Procedure: PCI — A loop recorder is implanted i all patients in both study groups to investigate:
  * Prevalence and severity of cardiac arrhythmias.
  * Effect on detected arrhythmia, in particular ventricular tachyarrhythmia, of optimal medical therapy vs. coronary revascularization by PCI.
  * Prevalence and severity of cardiac arrhythmias in CTO-patients with failed PCI.
  * Indication for prophylactic ICD implantation in CTO-patients treated conservatively or by PCI and after failed PCI.
  * Relation of arrhythmias to angina pectoris symptoms (CCS class), Quality of life questionnaire results and presence of myocardial reversible perfusion defects by CMRI.
  Other Names: Loop recorder
  Arms: Optimal Medical Treatment and PCI

SUMMARY:
In patients with a chronic total coronary occlusion (CTO ), clinically significant arrhythmia seems to be an important and a poorly investigated problem. The arrhythmia prevalence in an all-comer CTO-population is unknown, but in ICD-populations with ischemic heart disease, a CTO may be found in half of patients with life-threatening arrhythmia.The purpose of the CTO-ARRHYTHMIA study, is to investigate the incidence of clinically significant arrhythmias in CTO patients using an implantable loop recorder. Further, the investigators intend to identify predictors for arrhythmias as well as the impact on arrhythmia of optimized pharmacological treatment and revascularization in CTO patients.

DETAILED DESCRIPTION:
In angiographic materials, chronic total coronary occlusion (CTO) is present in approximately 15-25% of patients and in 25-50% of those with significant coronary disease. Until recently, because of low procedural success and increased risk of complications, PCI was a problematic treatment in these patients. The introduction of drug eluting stents and a variety of dedicated CTO devices combined with the evolution of specific CTO techniques have made revascularization by PCI a promising treatment.

In CTO patients, clinically significant arrhythmia seems to be an important and a poorly investigated problem. The arrhythmia prevalence in an all-comer CTO-population is unknown, but in ICD-populations with ischemic heart disease, a CTO may be found in half of patients with life-threatening arrhythmia. Further, in patients with ischemic heart disease receiving ICDs as primary prevention, presence of a CTO was an independent predictor of occurrence of ventricular arrhythmias, and in survivors of out-of-hospital cardiac arrest, the risk of ventricular arrhythmias was found to be increased in patients with a chronic total coronary occlusion. Nevertheless, the genesis of arrhythmia in CTO-patients is likely to be multifactorial. It has been documented, that ischemic heart disease patients who present with a chronic occlusion of at least one coronary artery are older and have additional risk factors such as hypertension, diabetes, lower left ventricular ejection fraction (LVEF) and more frequent myocardial infarction, i.e. a higher Chads2Vasc score (risk score for stroke in atrial fibrillation patients). Although LVEF is lower in patients with a chronic coronary occlusion, less than 1/3 are potential ICD candidates with an LVEF <35%. However, a recent study in consecutive post-AMI survivors documented the highest incidence of sudden cardiac death in patients with a relatively preserved LVEF.

The purpose of the CTO-ARRHYTHMIA study, is to investigate the incidence of clinically significant arrhythmias in CTO patients using an implantable loop recorder. Further, the investogators intend to identify predictors for arrhythmias as well as the impact on arrhythmia of optimized pharmacological treatment and revascularization in CTO patients. Here, CTO patients with failed PCI may be individuals with a particularly high risk of severe arrhythmias.

ELIGIBILITY:
Inclusion Criteria:

* ≥1 CTO lesion amenable to PCI.
* Stable or stabilized coronary artery disease.
* Angiographic/echocardiographic signs of reversible perfusion.
* CTO lesion in a coronary vessel supplying a significant myocardial territory (vessel diameter usually ≥3mm).

Exclusion Criteria:

* Expected survival <1 year.
* Patients with an indication of ICD due to EF < 35 or previous ventricular tachycardia.
* Patients with a cardiac device i.e. ICD, pacemaker or cardiac resynchronizing treatment device.
* Renal failure on dialysis.
* Lesions treated with PCI within one month.
* Indication for coronary artery bypass grafting (CABG). I.e. Two-or three vessel disease or left main disease and a syntax score >22.
* Significant valvular heart disease.
* Declined informed consent.
* Regarding CMRI: allergy to contrast medium, severe obesity, claustrophobia and certain metallic implants.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Rate of clinically significant arrhythmias | 1 year
  Rate og clinically significant arrhythmias in PCI versus medically only treated patients by loop recorder (table 1) and in patients with failed PCI.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Soegaard, DMSc, Study Chair — Co-PI
Locations (1):
- Aalborg university hospital, Aalborg, North Denmark, Denmark

IPD SHARING:
Plan to Share IPD: No
Data will be analyzed at site